CLINICAL TRIAL: NCT06598306
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-Tumor Activity of Subcutaneous Tarlatamab in Subjects With Extensive Stage Small Cell Lung Cancer (DeLLphi-308)
Brief Title: Subcutaneous Tarlatamab in Participants With Extensive Stage Small Cell Lung Cancer (DeLLphi-308)
Acronym: DeLLphi-308
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 20230298
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — AMG 757

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose Exploration (Experimental): Tarlatamab will be administered as a SC injection in Part 1.
  Interventions: Drug: Tarlatamab
- Part 2 Dose Expansion (Experimental): Following the selection of a SC dosing regimen in Part 1, tarlatamab will be administered in Part 2 at the dose deemed safe and tolerable in Part 1.
  Interventions: Drug: Tarlatamab
- Part 3 Alternative Dosing (Experimental): Following the selection of a SC dosing regimen from Part 1 that will be used in Part 2 dose expansion, Part 3 may open to test alternative dosing of SC tarlatamab.
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Administered by SC injection.
  Other Names: AMG 757; Imdelltra

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of subcutaneous (SC) tarlatamab.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years of age (or ≥ legal adult age within country if it is older than 18 years) at time of signing informed consent.
* Participants with histologically or cytologically confirmed ES-SCLC that progressed or recurred following at least one line of platinum-based anti-cancer therapy for SCLC.

Note: Participants with prior treatment for LS-SCLC should have also received another regimen for their recurrent, ES-SCLC disease.

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Participants must have adequate organ function (cardiac, pulmonary, kidney, and liver).
* Participants must be able to have SC injections administered in the abdomen.
* Participants without measurable disease or tumor tissue (fresh biopsy or archival) available may be permitted after discussion with and approval by Amgen Medical Monitor.

Exclusion Criteria:

* Participants that have received prior DLL3 targeted therapy.
* Participants with untreated or symptomatic brain metastases or those requiring therapy with steroids.
* Note: Participants with asymptomatic brain metastatic lesions are allowed following definitive treatment (Amgen Medical Monitor may approve untreated, asymptomatic brain metastasis if local therapy is not required per investigator judgment).
* Participants with leptomeningeal disease.
* Participants with baseline oxygen requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2030-03-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting toxicities (DLTs) | Up to day 21
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 24 months
Number of Participants with Changes in Vital Signs | Up to approximately 24 months
Number of Participants with Clinically Significant Changes in Clinical Laboratory Tests | Up to approximately 24 months

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Tarlatamab | Up to approximately 12 months
Serum Concentration Prior to Dosing (Ctrough) of Tarlatamab | Up to approximately 12 months
Time to Cmax (Tmax) of Tarlatamab | Up to approximately 12 months
Area Under the Concentration-time Curve (AUC) of Tarlatamab | Up to approximately 12 months
Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to approximately 24 months
Duration of Response (DOR) per RECIST 1.1 | Up to approximately 24 months
Time to Response (TTR) per RECIST 1.1 | Up to approximately 24 months
Progression-free Survival (PFS) per RECIST 1.1 | Up to approximately 24 months
Time to Progression per RECIST 1.1 | Up to approximately 24 months
Time to Subsequent Therapy | Up to approximately 24 months
Overall Survival (OS) | Up to approximately 24 months
Number of Participants with Anti-tarlatamab Antibody Formation | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (6):
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Illinois Chicago, Chicago, Illinois
  - Trinity Health Saint Joseph Mercy Ann Arbor, Ann Arbor, Michigan
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Australia (3):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China
- Germany (2):
  - Universitaetsklinikum Regensburg, Regensburg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Japan (2):
  - Okayama University Hospital, Okayama, Okayama-ken
  - Wakayama Medical University Hospital, Wakayama
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
- Spain (4):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (3):
  - Kantonsspital Graubuenden, Chur
  - Freiburg Spital, Fribourg
  - Kantonsspital Winterthur, Winterthur
- Turkey (Türkiye) (3):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Koc Universitesi Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com